CLINICAL TRIAL: NCT03261817
Title: Clinical and Brain Effects of Remote Web-based Adapted Physical Activity (e-APA) in Patients With Psychotic Disorders and Healthy Subjects: A Controlled, Multicenter Study
Brief Title: A Controlled Study With Remote Web-based Adapted Physical Activity (e-APA) in Psychotic Disorders
Acronym: PEPSYV@SI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No financial support
Sponsor: University Hospital, Caen (Other)
Collaborators: Centre Hospitalier du Rouvray (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-A00930-51
Record Dates: First submitted 2017-08-16; First posted 2017-08-25 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia; Physical Activity; Schizo Affective Disorder
Keywords: web; brain imaging; heart rate variability; circadian cycles; cognition; well-being; hippocampus; N acetyl aspartate; white matter; physical activity
MeSH Terms: conditions — Schizophrenia; Motor Activity; Psychotic Disorders | interventions — Exercise; Glutamyl Aminopeptidase

STUDY DESIGN:
Intervention Model Description: Randomization will be centralized and will be established for SCZ; Healthy Controls (HV) will be recruited by being matched to patients on age (according to 4 categories (18-25 years, 25-35 years, 35-50 years and> 50 years), gender and level of activity estimated by the self-administered questionnaire of Ricci and Gagnon.
  Randomization will be carried out in two arms:
  * interventional (adapted physical activity APA)
  * control (health education program)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- APA in patients (Experimental): patients receiving physical activity (APA) by web during 16 weeks with 2 sessions a week
  Interventions: Behavioral: Physical activity (APA)
- HE in patients (Sham Comparator): patients receiving Health education program (HE) by web during 16 weeks with 2 sessions a week
  Interventions: Behavioral: Health Education program (HE)
- APA in healthy volunteer controls (Active Comparator): Healthy volunteers receiving physical activity (APA) by web during 16 weeks with 2 sessions a week
  Interventions: Behavioral: Physical activity (APA)
- HE in healthy volunteer controls (Sham Comparator): Healthy volunteers receiving Health education program (HE) by web during 16 weeks with 2 sessions a week
  Interventions: Behavioral: Health Education program (HE)

INTERVENTIONS:
Behavioral: Physical activity (APA) — 2 sessions a week of 1 hour during 16 weeks. APA exercises by web will be aerobic type associated with muscle toning program; Activities will combine relaxation techniques, body expression and muscle relaxation (yoga, stretching, relaxation, step etc ...).
  The intensity of the activities will be individualized for each participant according to his/her physical condition
  Arms: APA in healthy volunteer controls; APA in patients
Behavioral: Health Education program (HE) — 2 sessions a week of 1 hour during 16 weeks HE by web will be delivered and was composed of information on the main mental disorders, the benefits of physical activity, healthy lifestyle (dietary balance, sleep cycle, stress management), alcohol, drug, tobacco and cardiovascular risk factors
  Arms: HE in healthy volunteer controls; HE in patients

SUMMARY:
In this study, an APA program by web (e-APA) will be offered to two groups of participants (21 patients and 21 healthy volunteers (HV)) in remote video (use of the SAPATIC (Santé Activités Physiques Adaptées utilisant les Technologies de l'Information et de la Communication) platform developed by the company V@SI). At the same time, two control groups, a group of 21 patients and a group of 21 HV will undergo an health education program (HE) through the collaborative SAPATIC health platform of V@Si and will constitute the control groups. The content of the APA sessions will be administered by V@Si. This program offers content aimed to improve aerobic capacity and muscular strength while relying on the motivation of the participants

DETAILED DESCRIPTION:
The main objective is to demonstrate that APA can improve cerebral plasticity in patients with schizophrenic or schizoaffective disorders (SCZ), reflected by an increase in the overall volume of hippocampus.

The secondary objectives will also be to assess the impact of APA on the SCZ compared to the HV:

1. on other cerebral variables (changes in the different subregions of the hippocampus (Cornu Ammonis (CA: CA1,CA2-3-4), subiculum and dentate gyrus), cortical thickness, N-acetyl aspartate (NAA) and glutamate as well as changes in the white matter through the diffusion markers (fractional anisotropy, radial diffusivity and mean diffusivity in the frontomedial-hippocampal fibers) and cerebral irrigation
2. on physiological variables (neuromuscular, cardiovascular (heart rate variability) and aerobic)
3. on cognitive variables by measuring working memory, episodic memory, attentional and executive functions
4. on circadian rhythms (temperature, actimetry and wake-sleep cycle)
5. on the clinical status of patients (severity of symptoms, quality of life, level of activity and physical abilities).
6. on biological variables (fasting glucose, triglycerides, total cholesterol, High-density lipoprotein cholesterol (HDLc), Low-density lipoprotein cholesterol (LDLc)

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Be over 18 years of age and under 60 years of age
* with schizophrenia or schizoaffective disorder according to DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, 4th edition) criteria established with a semi-structured interview (Mini International Neuropsychiatric Interview, French version 5.0.0).
* The possibility of receiving each of the 2 interventions (APA or HE)
* No change in psychotropic drugs (antidepressants, antipsychotics or mood regulators) during the 2 months prior to inclusion for patients.
* Collecting the signature of informed consent.
* The need to be affiliated to a medical welfare
* The agreement of the guardian or trustee in case of a protected major

Healthy Volunteers:

* between 18 and 60 years old
* The possibility of receiving each of the 2 interventions (APA or HE)
* Collecting the signature of informed consent.
* The need to be affiliated to a medical welfare

Exclusion Criteria:

Patients with only one of the non-inclusion criteria may not be eligible to participate in the research. These criteria are:

* Age under 18 or over 60 years old
* Pregnancy
* The inclusion of the patient in another biomedical research protocol (during the present study)
* Patients with progressive neurological disease
* Patients with contraindications to MRI (including electronic or metal implants)
* Patients who refused to wear earplugs during the MRI examination
* Patients with a physical contraindication to physical activity (moderate to severe heart failure, severe valvular disease, unstable coronary disease, acute pulmonary embolism or untreated deep venous thrombosis, uncontrolled hypertension, pulmonary arterial hypertension, treaty)
* Neuromuscular pathologies, severe sensory and / or motor neuropathy
* Rheumatic and articular pathologies; Rheumatologic / orthopedic problems or bone lesions at risk of fracture contraindicating physical activity
* History of stroke or myocardial infarction less than 6 months old at the selection visit

Healthy Volunteers

Participants with only one of the non-inclusion criteria may not be eligible to participate in the research. These criteria are:

* Age under 18 or over 60 years old
* Pregnancy
* Inclusion of the participant in another biomedical research protocol (during this study)
* Participants with progressive neurological disease
* Participants with a contraindication to MRI (including electronic or metal implants)
* Participants refused to wear ear plugs during the MRI examination
* Participants with life-long schizophrenia or schizoaffective disorder according to the DSM-IV criteria established with a semi-structured interview (Mini International Neuropsychiatric Interview, MINI; French version 5.0.0).
* Presence of cardiovascular pathologies contraindicating physical activity (moderate to severe heart failure, severe valvular disease, unstable coronary disease, acute pulmonary embolism or untreated deep venous thrombosis, uncontrolled hypertension, pulmonary arterial hypertension, rhythm disorder untreated)
* Neuromuscular pathologies, severe sensory and / or motor neuropathy
* Rheumatic and articular diseases, rheumatological / orthopedic problems or fracture risk bone lesions
* History of stroke or myocardial infarction less than 6 months old at the selection visit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
hippocampal volumes | at Day 127 +/- 8 days or after 10 sessions of APA if premature cessation of treatment
  The primary endpoint is the right and left hippocampal volumes

SECONDARY OUTCOMES:
Cerebral variables | at Day 127 +/- 8 days or after 10 sessions of APA if premature cessation of treatment
  changes in the different subregions of the hippocampus (CA1, CA2-3-4, subiculum and dentate gyrus, cortical thickness, N-acetyl aspartate (NAA) and glutamate as well as changes in the white matter through the diffusion markers (fractional anisotropy, radial diffusivity and mean diffusivity in the frontomedial-hippocampal fibers) and cerebral irrigation
Physiological variables | at Day 127 +/- 8 days or after 10 sessions of APA if premature cessation of treatment
  neuromuscular, cardiovascular (heart rate variability) and aerobic (VO2)
Circadian rhythms | at Day 127 +/- 8 days or after 10 sessions of APA if premature cessation of treatment
  temperature, actimetry and wake-sleep cycle
Clinical status | at Day 127 +/- 8 days or after 10 sessions of APA if premature cessation of treatment
  severity of symptoms, quality of life, level of activity and physical abilities
Biological variables | at Day 127 +/- 8 days or after 10 sessions of APA if premature cessation of treatment
  fasting glucose, triglycerides, total cholesterol, HDLc, LDLc

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leroux E, Trehout M, Reboursiere E, de Flores R, Morello R, Guillin O, Quarck G, Dollfus S. Effects of web-based adapted physical activity on hippocampal plasticity, cardiorespiratory fitness, symptoms, and cardiometabolic markers in patients with schizophrenia: a randomized, controlled study. Eur Arch Psychiatry Clin Neurosci. 2024 Sep;274(6):1245-1263. doi: 10.1007/s00406-024-01818-8. Epub 2024 May 13. PMID 38740618
- [Derived] Trehout M, Leroux E, Bigot L, Jego S, Leconte P, Reboursiere E, Morello R, Chapon PA, Herbinet A, Quarck G, Dollfus S. A web-based adapted physical activity program (e-APA) versus health education program (e-HE) in patients with schizophrenia and healthy volunteers: study protocol for a randomized controlled trial (PEPSY V@Si). Eur Arch Psychiatry Clin Neurosci. 2021 Mar;271(2):325-337. doi: 10.1007/s00406-020-01140-z. Epub 2020 May 26. PMID 32458107